CLINICAL TRIAL: NCT02338011
Title: Gefitinib Alone or With Concomitant Whole Brain Radiotherapy for Patients Harboring an EGFR Mutation With Multiple Brain Metastases From Non-Small-cell Lung Cancer: a Phase II/III Randomized Controlled Trial
Brief Title: Comparator-Controlled Study for EGFR(+) Patients With Multiple BMs From NSCLC (BROKE) (EGFR-epidermal Growth Factor Receptor;BM-brain Metastases)
Acronym: EGFR
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Liyan Jiang, Director of Department of Respiratory, Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiChest Hospital
Record Dates: First submitted 2014-12-23; First posted 2015-01-14 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Non-Small Cell Lung Cancer; Brain Metastases; EGFR Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gefitinib alone (Experimental): Patients harboring an EGFR mutation with multiple BM from NSCLC will receive Gefitinib 250mg per day until progression of disease.
  Interventions: Drug: Gefitinib
- Gefitinib concurrent WBRT (Experimental): Patients harboring an EGFR mutation with multiple BM from NSCLC will receive Gefitinib concurrent WBRT until progression of disease.Gefitinib was given 250mg per day. WBRT was delivered in 3.0 Gy fractions once per day 5 days per week to a total dose of 30Gy (10 fractions).
  Interventions: Drug: Gefitinib; Radiation: WBRT

INTERVENTIONS:
Drug: Gefitinib — Gefitinib was given 250mg per day. Dose reduction was allowed for intolerable adverse effects such as rash(grade 4)、diarrhea(grade 3-4) or non hematological toxicity(grade 3-4) from 250mg per day to 250mg every other day then to 250mg every three days if needed.
  Other Names: Iressa
Radiation: WBRT — WBRT was delivered in 3.0 Gy fractions once per day 5 days per week to a total dose of 30Gy (10 fractions).
  Arms: Gefitinib concurrent WBRT

SUMMARY:
1. Compare the effect and safety of gefitinib alone with gefitinib plus concomitant WBRT(whole-brain radiotherapy ) in treatment of NSCLC patients harboring an EGFR mutation with multiple BM.
2. Verify the failure pattern of NSCLC patients harboring an EGFR mutation with multiple BM.
3. Explore the rescuable therapy after progression of disease.

DETAILED DESCRIPTION:
All patients will be randomized to receive gefitinib or gefitinib concurrent WBRT until progression of disease. Gefitinib concurrent WBRT, patients were given gefitinib 250mg per day concurrently with WBRT(whole-brain radiotherapy ). Dose reduction was allowed for intolerable adverse effects such as rash(grade 4)、diarrhea(grade 3-4) or non hematological toxicity(grade 3-4) from 250mg per day to 250mg every other day then to 250mg every three days if needed. WBRT was delivered in 3.0 Gy(Gray)fractions once per day 5 days per week to a total dose of 30Gy (10 fractions). Radiation was delivered as opposed lateral 6-MV(Micro Voltage) beams with Varian linear accelerator.

ELIGIBILITY:
Inclusion Criteria:

* years of age or older
* ECOG score ≤ 2
* Recursive Partitioning Analysis(RPA) Class I-II;
* The pathological diagnosis of primary non-small cell lung cancer and detection of pulmonary primary ARMs;
* Sequencing EGFR mutation(primary lesion or metastases,exon 19 deletions or exon 21 L858R (EGFR mutation in exon 21, L858R point mutation) mutations;
* Enhanced MRI showed brain metastases ≥ 4;
* 1 or 2 line treatment revealed failure;

  * No use of EGFR-TKIs(Tyrosine kinase inhibitors) previously；
  * No treatment for BM previously,including WBRT、SRS、surgery or experimental therapy;
  * Expected survival period over 3 months;
  * Two weeks before randomization, organs function in patients with meet the following criteria:

    * bone marrow:HB(hemoglobin) ≥ 90g/L, neutrophil≥ 1.5 × 109/L and platelet ≥ 100 × 109/L;
    * liver function:total bilirubin ≤ 1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal;
    * renal function:more than 1.5 times the upper limit of normal serum creatinine or creatinine clearance rate ≥ 60 ml/min;
    * Urine dipstick testing the proteinuria < 1+; if the urine dipstick test value, 1+, is 24 hours total urine protein must < 500mg;
    * blood glucose:normal range,DM(diabetes mellitus) patients are under treatment and have a stable state;
  * Can understand and consent

Exclusion Criteria:

* Patients have been treated with brain radiation or surgery of BM;
* Prior of EGFR-TKIs；
* Mixed with small cell lung cancer patients with components;
* Wild-type of EGFR;
* Unable to tolerate MRI scanning;
* Post 2 line treated patients;
* Brain meninges metastases or incorporate with brain meninges metastases;
* 5 years before other cancers except NSCLC treatment in patients with the start of the study (except for simple operation resection and there are at least 5 consecutive years disease free survival, has been cured of cervical carcinoma in situ, has cured the base cell cancer and bladder epithelial tumor);
* Before entering the group 4 weeks received any other investigational drugs;
* Incorporate with local symptoms（hemiplegic paralysis、anepia、nystagmus、ataxia.et);
* Pregnancy or lactation female;
* Allergic to EGFR-TKIs or any components;
* Patients were not permitted to receive the following drugs: phenytoin, carbamazepine, rifampicin, phenobarbital or itraconazole because of their potential to affect the metabolism of EGFR-TKIs and reduce its plasma concentration. Patients were not permitted to receive oral medicine such as CoumadinTM、Warfarin. If anticoagulant therapy is needed,low molecular heparin is suggested to instead of Coumarin drugs;
* Organs function in patients with meet the following criteria:

  * Diagnose with interstitial lung disease、drug induced interstitial disease、hormone dependent radiation pneumonia previously,et al;
  * Any unstable system diseases: including active infection, moderate to severe chronic obstructive pulmonary disease, uncontrolled hypertension, unstable angina pectoris, congestive heart failure, within the last 6 months of the onset of myocardial infarction, need serious mental disorder drug treatment, liver, kidney or metabolic diseases; mental / spiritual diseases such as Alzheimer's disease;
  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption or active peptic ulcer;
  * With immunodeficiency disease, or suffer from other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
  * Known human immunodeficiency virus (HIV) infection;
  * Without full control of ocular inflammation or eye infections, or any may cause the eye disease situation;
* Any disease, metabolic disorders, or physical examination or laboratory suspicion or treatment of complications in patients at high risk of drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 12-14 months
  Compare the progression free survival(PFS) and safety in two arms,including intracranial PFS、extracranial PFS and overall PFS.

SECONDARY OUTCOMES:
Overall survival | 3 years
Disease Progression Classification | 3 years
  intracranial or extracranial site
Health-related quality of life | 3 years
  measured by ECGO(Eastern Cooperative Oncology Group) PS (Performance Status)
Mental Status | 3 years
  measured by scale of MMSE( Mini Mental Status Examination)

CONTACTS AND LOCATIONS:
Overall Officials: Liyan JIang, M.D,Ph.D., Study Director — Department of Respiratory, Shanghai Chest Hospital,Shanghai JIaotong University
Locations (1):
- Varian linear accelerato, Shanghai, Shanghai Municipality, China